CLINICAL TRIAL: NCT07375017
Title: Evaluation of the Safety and Effectiveness of easyEndo™ Powered Single Use Powered Endoscopic Staplers and Cartridges in Laparoscopic Bariatric Procedures: an Observational, Post Market Study
Brief Title: easyEndoTM Powered Stapler Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-BS-QA
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- easyEndo™ Powered Single Use Powered Endoscopic Staplers and Cartridges (Experimental): The easyEndoTM Powered Single Use Powered Endoscopic Staplers and Cartridges, which used together, are intended for transection, resection, and/or creation of anastomoses. The instruments have application in multiple open or minimally invasive general abdominal, gynecologic, thoracic, and pediatric surgical procedures.
  Interventions: Device: laparoscopic bariatric surgery

INTERVENTIONS:
Device: laparoscopic bariatric surgery — laparoscopic bariatric surgery using easyEndo™ Powered Single Use Powered Endoscopic Staplers and Cartridges

SUMMARY:
The goal of this Observational, retrospective, uncontrolled is to evaluate the safety and performance of the easyEndo™ Powered Single Use Powered Endoscopic Staplers and Cartridges from EziSurg Medical used in laparoscopic bariatric surgery.. The main question it aims to answer the safety and performance of the device

ELIGIBILITY:
Inclusion Criteria:

* Patients have undergone laparoscopic bariatric surgery.
* The operation involves the application of easyEndo™ Powered Staplers and Cartridges for tissue cutting and suturing.

Exclusion Criteria:

* Pregnancy.
* Emergency operation (such as acute intestinal obstruction and gastrointestinal perforation).
* Assessed by the investigator, whose condition is poor and cannot tolerate the surgery.
* History of gastrointestinal surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
stapling success rate | Perioperative/Periprocedural
  no leakage intra-operation and post-operation

SECONDARY OUTCOMES:
postoperative complications | Perioperative/Periprocedural
  postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- The Masters Medical Center, Doha, Doha Municipality, Qatar

IPD SHARING:
Plan to Share IPD: No